CLINICAL TRIAL: NCT01298687
Title: Divided Dose of TRAVATAN®
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-10-081
Record Dates: First submitted 2011-02-16; First posted 2011-02-18 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2014-07

CONDITIONS: Open-angle Glaucoma; Ocular Hypertension
Keywords: open-angle glaucoma; ocular hypertension; divided dose
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Travoprost

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Trav 0.00013% (Experimental): Travoprost Ophthalmic Solution, 0.00013%, 1 drop administered in each eye 12 times per day at 2-hour intervals for 5 days
  Interventions: Drug: Travoprost Ophthalmic Solution, 0.00013%
- Trav 0.00033% (Experimental): Travoprost Ophthalmic Solution, 0.00033%, 1 drop administered in each eye 12 times per day at 2-hour intervals for 5 days
  Interventions: Drug: Travoprost Ophthalmic Solution, 0.00033%
- Trav 0.001% (Experimental): Travoprost Ophthalmic Solution, 0.001%, 1 drop administered in each eye 12 times per day at 2-hour intervals for 5 days
  Interventions: Drug: Travoprost Ophthalmic Solution, 0.001%
- Trav 0.00267% (Experimental): Travoprost Ophthalmic Solution, 0.00267%, 1 drop administered in each eye 12 times per day at 2-hour intervals for 5 days
  Interventions: Drug: Travoprost Ophthalmic Solution, 0.00267%
- TRAVATAN (Active Comparator): Travoprost Ophthalmic Solution, 0.004%, 1 drop administered in each eye at 8 pm for 5 days, with 1 drop of vehicle administered at all other timepoints (2-hour intervals)
  Interventions: Drug: Travoprost Ophthalmic Solution, 0.004%
- Vehicle (Placebo Comparator): Travoprost vehicle, 1 drop administered in each eye 12 times per day at 2-hour intervals for 5 days
  Interventions: Drug: Travoprost Vehicle

INTERVENTIONS:
Drug: Travoprost Ophthalmic Solution, 0.00013% — Cumulative daily dose is below the travoprost ophthalmic solution, 0.004% once daily dose
  Arms: Trav 0.00013%
Drug: Travoprost Ophthalmic Solution, 0.00033% — Cumulative daily dose equals the travoprost ophthalmic solution, 0.004% once daily dose
  Arms: Trav 0.00033%
Drug: Travoprost Ophthalmic Solution, 0.001% — Cumulative daily dose is above the travoprost ophthalmic solution, 0.004% once daily dose
  Arms: Trav 0.001%
Drug: Travoprost Ophthalmic Solution, 0.00267% — Cumulative daily dose is above the travoprost ophthalmic solution, 0.004% once daily dose
  Arms: Trav 0.00267%
Drug: Travoprost Ophthalmic Solution, 0.004%
  Other Names: TRAVATAN®
  Arms: TRAVATAN
Drug: Travoprost Vehicle — Inactive ingredients used as an active comparator
  Arms: Vehicle

SUMMARY:
The purpose of this study is to compare the incremental dosing of travoprost ophthalmic solution versus once a day dosing of TRAVATAN® in lowering intraocular pressure (IOP) in patients with open-angle glaucoma (OAG) or ocular hypertension (OHT).

ELIGIBILITY:
Inclusion Criteria:

* Patients with open-angle glaucoma or ocular hypertension who meet the following IOP criteria:

  1. Mean IOP ≥ 24 mmHg in at least 1 eye, with the same eye qualifying at 8 AM at both Day 0 and Day 1;
  2. Mean IOP ≤ 36 mmHg in both eyes at all time points on Day 0 and Day 1.
* Must sign an informed consent form.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Females of childbearing potential who are pregnant, test positive on urine pregnancy test at the Screening Visit, intend to become pregnant during the study period, are breast-feeding, or are not using highly effective birth control measures.
* Current or history of ocular inflammation or infection in either eye within the past 3 months.
* Corneal thickness greater than 620 µm as determined by pachymetry in either eye.
* Severe visual field loss.
* Cup to disc ratio greater than 0.8 in either eye.
* Intraocular surgery within the past 6 months in either eye.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2011-02; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
24-hour Area Under the Curve (AUC) in IOP Reduction | Day 5

CONTACTS AND LOCATIONS:
Overall Officials: Matt Walker, PhD, Study Director — Alcon Research